CLINICAL TRIAL: NCT03016559
Title: Effect of Releasing Quadratus Lumborum Muscle on Angles of Hip Joint in Asymptomatic Individuals
Brief Title: Effect of Releasing Quadratus Lumborum Muscle on Hip Joint Range of Motion in Asymptomatic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MahidolU_Wunpen2
Record Dates: First submitted 2017-01-08; First posted 2017-01-10 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Muscle
Keywords: releasing muscle; quadratus lumborum; hip angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- releasing muscle (Other): The physical therapist placed thumbs on the quadratus lumborum to release muscle.
  Interventions: Other: releasing muscle

INTERVENTIONS:
Other: releasing muscle — At baseline, hip and knee angles were measured. The quadratus lumborum muscle was released. After that, the hip and knee angles were re-measured.

SUMMARY:
The purpose of this study are to compare angles of hip joint between before and after releasing quadratus lumborum muscle.

DETAILED DESCRIPTION:
The 1st physical therapist performed the modified Thomas test position. The participant was asked to lie supine over the edge of the couch. The participant hold one knee to the chest tightly while the other knee was bent over the end of the couch. The 2nd physical therapist measured angles of hip and knee using a standard goniometer at baseline. The quadratus lumborum muscle was released. Then the same measurement was repeated.

ELIGIBILITY:
Inclusion Criteria:

1. asymptomatic male and female volunteers
2. age 18-65 years

Exclusion Criteria:

1. having musculoskeletal symptoms (e.g. fibromyalgia, pain at any regions, instability of lower extremities caused by ligamentous injury, injury or trauma to lower extremities), endocrine disease, rheumatoid arthritis
2. taking muscle relaxant or pain killer within 1 day prior to data collection
3. having past history of low back and hip surgery
4. pregnancy
5. having menstruation on data collection day
6. having joint deformities (e.g. knock knee, bow leg)

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Hip abduction angle | 5 minutes
  Range of motion (ROM) of hip abduction

SECONDARY OUTCOMES:
Hip flexion angle | 5 minutes
  Range of motion (ROM) of hip flexion

OTHER OUTCOMES:
Knee flexion angle | 5 minutes
  Range of motion (ROM) of knee flexion

CONTACTS AND LOCATIONS:
Overall Officials: Chompunoot Suwanasri, MSc, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jairakdee Y, Chansirinukor W, Sitti T. Effect of releasing quadratus lumborum muscle on hip and knee muscle length in asymptomatic individuals. J Bodyw Mov Ther. 2021 Apr;26:542-547. doi: 10.1016/j.jbmt.2020.11.008. Epub 2020 Nov 7. PMID 33992295